CLINICAL TRIAL: NCT02153892
Title: Clinical Protocol - A Feasibility Study Using the AccuCinch® System in the Left Ventricular Reshaping of the Mitral Apparatus to Reduce Functional Mitral Regurgitation and Improve Left Ventricular Function
Brief Title: Feasibility of the AccuCinch® System for Left Ventricular Reshaping of the Mitral Apparatus to Reduce Functional Mitral Regurgitation and Improve Left Ventricular Function
Acronym: LVRECOVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ancora Heart, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3870
Record Dates: First submitted 2014-05-28; First posted 2014-06-03 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Severe Functional Mitral Regurgitation and Heart Failure
Keywords: Functional Mitral Regurgitation; Heart Failure; Ventricular Reshaping
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Multi-center, prospective, single-arm study (Other): To assess the safety and performance of the GDS Accucinch System when used percutaneously to reduce functional mitral regurgitation.
  Interventions: Device: GDS Accucinch System

INTERVENTIONS:
Device: GDS Accucinch System — Percutaneous Coronary Intervention

SUMMARY:
To assess the safety and performance of the GDS Accucinch System when used percutaneously to reduce functional mitral regurgitation.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Subjects with severe symptomatic functional mitral regurgitation of ≥ 3+ secondary to left ventricular (LV) remodeling and/or annular remodeling, as measured in accordance with the current ASE guidelines and suitable for treatment in accordance with the current AHA/ACC guidelines:

  * Left ventricular ejection fraction (LVEF) ≥ 20% and ≤ 40%
  * Stable cardiac medical regimen for heart failure for at least 1 month
  * Stable NYHA Classification (Class III and above) for at least 1 month
* The subject has been informed of the nature of the study, agrees to its provisions, including the possibility of conversion to surgery, and has provided written informed consent.

Exclusion Criteria:

Candidates will be excluded from the study if any of the following conditions are present:

* Myocardial infarction within 90 days of the intended treatment with the device
* Prior surgical, transcatheter, or percutaneous mitral valve intervention or mitral valve prosthesis
* Subject has untreated coronary artery disease, which in the opinion of the treating physician and/or heart team, is clinically significant and requires revascularization
* Non-ambulatory NYHA Class IV symptoms of heart failure or subjects in cardiogenic shock or with hemodynamic instability requiring IV inotropic support or mechanical support devices
* Subject has the need for emergent surgery for any reason
* Subjects in whom sufficient quality of echocardiography (TTE and TEE) cannot be obtained
* Echocardiography evidence of primary mitral valve disease causing MR or MS;
* Moderate to severe pulmonary hypertension (PA systolic pressure ≥ 80 mm Hg) as assessed by echocardiography
* Evidence of mitral valve stenosis with an estimated valve area less than 3.5 cm2
* Mitral valve pathology that would prevent adequate function of the GDS Accucinch System
* Subject is on dialysis or estimated GFR < 30mL/min/1.73m2 (Cockcroft-Gault Formula)d d Israni AK, et al. Laboratory Assessment of Kidney Disease, in Brenner and Rector's The Kidney, 9th ed. chapter 25
* Greater than mild mitral annular calcification observed by fluoroscopy
* Presence of aortic valve prosthesis
* Moderate to severe aortic valve stenosis or calcification observed by echocardiography or fluoroscopy
* Severe aortic arch calcification or mobile aortic atheroma observed by echocardiography or fluoroscopy
* Active bacterial endocarditis or active sepsis
* History of bleeding diathesis or coagulopathy
* History of stroke within the prior 6 months
* Subjects in whom anticoagulation is contraindicated
* Any clinical evidence that the investigator feels would place the subject at increased risk with the placement of the device
* Concurrent medical condition with a life expectancy of less than 12 months
* Currently participating in another investigational drug or device study that has not reached its primary endpoint
* Co-morbid conditions that place the subject at an unacceptable surgical risk (e.g. severe chronic obstructive pulmonary disease, hepatic failure, immunological abnormalities, and hematological abnormalities)
* Subject with indication for concomitant surgery such as coronary artery bypass graft (CABG), aortic valve reconstruction or replacement, left ventricular remodeling surgery and congenital repair
* Any cardiac resynchronization therapy within the last 9 months prior to treatment
* Subject on high dose steroids or immunosuppressant therapy
* Current problems with substance abuse (e.g. alcohol, illegal drugs, etc.)
* Female subjects who are pregnant, lactating, or planning pregnancy within next the 36 months. Note: Childbearing age should be instructed to use safe contraception during their participation in this study.
* Subjects who are unable or unwilling to comply with the follow-up schedule and requirements
* Subject has known hypersensitivity to contrast agents that cannot be adequately pre-medicated or has known hypersensitivity to study required medications, to nickel, or to polyurethanes
* Femoral artery lumen diameter of < 5.5 mm, or severe ilio-femoral tortuosity or calcification that would prevent safe placement of the 16Fr introducer sheath

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-08; Primary Completion 2015-10 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Procedural Success | 72 hours post-procedure
  Successful use and implantation of an Accucinch System without Major Adverse Events (MAE) defined as the occurrence of any of the following: All-cause mortality, Device and/or procedure-related death; Peri-procedural myocardial infarction (MI) < or equal to 72 hrs after index procedure; Major stroke; Urgent or emergent conversion to surgery or repeat procedure (surgical or interventional therapy) for mitral valve or heart failure related deterioration; Left ventricular perforation; Major vascular complications; Major bleeding (including cardiac tamponade)
Device Success | 24 hours post-procedure
  Successful vascular access, delivery, and retrieval of the delivery system; Ability to establish access to the sub-annular groove, to deploy the Anchors, and the Anchor Links, to apply tension to the Cinch Cable, to reshape the mitral annulus, to deploy the Lock, and to cut the Cinch Cable; Intended performance of the Accucinch System measured by TTE acutely post-cinch with a reduction of MR by at least one grade
Clinical Safety Measures | 7 day post procedure
  Defined as freedom from MAE at discharge or 7 days post-procedure, whichever comes first; Safety measures will be reviewed and adjudicated by an independent clinical events committee (CEC); Echocardiographic measures will be assessed by an independent echocardiography core laboratory

SECONDARY OUTCOMES:
Clinical Measure | 30 day post-procedure
  NYHA Class improvement of at lease one score from baseline
Echocardiographic Measures - Composite | 30 days post-procedure
  Mitral Valve Measures: One grade reduction in MR (e.g. 3+ to 2+), or; Reduction in PISA EROA at least 25% from baseline, or; Reduction in Regurgitant Volume at least 25% Left Ventricular Measures: Reduction in Left Ventricular size (Left Ventricular End Diastolic Dimension - LVEDD) at least 5% from baseline, or: Reduction in Left Ventricular volume (Left Ventricular End Diastolic Volume -LVEDV) at least 5%, or Increase in ejection fraction (LVEF) at least 10% from baseline Left Atrial Measures: Left atrial volume index (biplane area-length method). The above echocardiographic measures will be assessed by an independent core laboratory
Clinical Measure | 30 day post-procedure
  6-minute walk test compared to baseline
Clinical Measure | 30 day post-procedure
  Quality of Life (KCCQ Questionnaire) compared to baseline

OTHER OUTCOMES:
Additional Measures - Composite | Collected at baseline, peri- and post-procedure, discharge or 7-days (whichever comes first) 30-day, 3, 6, and 12 months and at 2 and 3 years post procedure
  Safety measures (adjudicated by an independent Clinical Events Committee): Mortality: all-cause, cardiovascular, and non-cardiovascular; Spontaneous Myocardial Infarction (>72 hrs post-index procedure); Major and life-threatening bleeding; Major stroke: disabling and non-disabling; Major vascular complication (access site, non-access site); Acute Kidney Injury (< or equal to 72 hrs post-procedure): based on the modified RIFLE Stage 3 (including renal replacement therapy), Stage 2, and Stage 1; Failure of current therapy for functional mitral regurgitation requiring re-hospitalization or prolonged hospitalization for FMR-related symptoms and worsening heart failure with NYHA class III or IV, or requiring conversion to surgery; Anchor(s) migration or Anchor(s) dislocation (as assessed by fluoroscopic images or CT) (when applicable)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zapien, Study Director — Ancora Heart, Inc.
Locations (1):
- Monash Health, Melbourne, Victoria, Australia